CLINICAL TRIAL: NCT01470456
Title: An Open Label, Multicenter Phase II Study of Intravenous SAR3419, an Anti-CD19 Antibody-Maytansine Conjugate, in Combination With Rituximab in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphomas
Brief Title: Combination of SAR3419 and Rituximab in Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD12333; 2011-002865-39; U1111-1120-0315 (Other: UTN)
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — coltuximab ravtansine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SAR3419 + Rituximab (Experimental): Combined therapy will be administered intravenously for 8 doses in the absence of unacceptable toxicity, disease progression or withdrawal of consent.
  Interventions: Drug: SAR3419; Drug: rituximab

INTERVENTIONS:
Drug: SAR3419 — Pharmaceutical form:solution for infusion Route of administration: Intravenous
Drug: rituximab — Pharmaceutical form:solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

Participants Achieving an Objective Response Rate (Cheson 2007)

Secondary Objectives:

* Progression Free Survival
* Overall Survival
* Response Duration

DETAILED DESCRIPTION:
* The screening period = up to 4 weeks prior to the first administration of combined therapy
* The treatment period = 3 months of combined therapy. A safety follow-up of 42 to 49 days after the last dose of treatment is planned for all patients.
* The follow-up period: Patients who are not progressing at the end of study treatment will be followed until progression or initiation of another anti-lymphoma therapy. All patients will be followed for two years to evaluate survival.

ELIGIBILITY:
Inclusion criteria:

* Histological diagnosis of Diffuse Large B-Cell Lymphoma (DLBCL)
* Relapsed or refractory after at least one standard treatment including rituximab
* CD19 and CD20 positive disease

Exclusion criteria:

* No bi-dimensionally measurable lesion by CT scan (defined as presence of at least one tumor mass measuring >1.5 x 1.5 cm)
* The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving an Objective Response Rate | 18 weeks

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Up to 6 months
Response Duration -Time | Up to 24 months after the first infusion of the last patient
Progression Free Survival -Time | Up to 24 months after the first infusion of the last patient
Overall survival -Time | Up to 24 months after the first infusion of the last patient

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- Investigational Site Number 040002, Graz, Austria
- France (11):
  - Investigational Site Number 250004, Créteil
  - Investigational Site Number 250009, Dijon
  - Investigational Site Number 250006, Lille
  - Investigational Site Number 250011, Marseille
  - Investigational Site Number 250010, Montpellier
  - Investigational Site Number 250008, Nantes
  - Investigational Site Number 250007, Paris
  - Investigational Site Number 250001, Pierre-Bénite
  - Investigational Site Number 250005, Rennes
  - Investigational Site Number 250003, Rouen
  - Investigational Site Number 250002, Villejuif
- Investigational Site Number 578001, Oslo, Norway